CLINICAL TRIAL: NCT00269607
Title: Naltrexone Implants as an Aid in Preventing Relapse Following Inpatient Treatment for Opioid Addiction.
Brief Title: Naltrexone Implants as Relapse Prevention
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment difficulties. Reframed as pilot study
Sponsor: University of Oslo (Other)
Responsible Party: University of Oslo, Institute of Psychiatry, Professor Edvard Hauff, Institute of Psychiatry, University of Oslo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11899
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2005-12

CONDITIONS: Opioid Dependency
Keywords: Substance abuse; Treatment; Relapse prevention; opioid antagonist
MeSH Terms: conditions — Substance-Related Disorders

INTERVENTIONS:
Drug: Implantation of naltrexone implants

SUMMARY:
The purpose of this clinical trial is to study the efficacy and safety of naltrexone implants as relapse prevention for patients that are completing treatment for opiate addiction in inpatient (or similarly controlled) settings. Participants in the naltrexone experimental group are prematched in a pairwise fashion with other patients who do not want a naltrexone implant during the first six months after ending inpatient treatment, but who reiceive treatment as usual (TAU) from the Norwegian healthcare system.

The hypotheses are that quality of life, depression, opioid use, will be significantly better in the naltrexone group compared to the non at 6-, 12-, and 18-month follow-up.

We also hypothesize that the implants can prevent death from opioid overdose up to 6 months after commenced treatment.

ELIGIBILITY:
Inclusion Criteria:

* soon to complete inpatient treatment for opioid addiction
* living in southern Norway

Exclusion Criteria:

* psychosis / major depression, currently not treated
* pregnancy
* liver enzymes: ASAT or ALAT > threefold above upper boundary
* maintenance treatment with methadone or buprenorphine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: drug use at 6(12/18)months by self report, hair analysis; days in work or education, number of drug-free friends at 6 (12/18)months by self report

SECONDARY OUTCOMES:
Secondary Outcomes: depression at 6(12/18)months by BDI and Hopkins SCL-25; quality of life at 6(12/18)months by EuropASI

CONTACTS AND LOCATIONS:
Overall Officials: Helge Waal, professor, Study Director — Unit for addiction medicine, Institute of psychiatry, University of Oslo

REFERENCES:
- [Derived] Kunoe N, Lobmaier P, Vederhus JK, Hjerkinn B, Gossop M, Hegstad S, Kristensen O, Waal H. Challenges to antagonist blockade during sustained-release naltrexone treatment. Addiction. 2010 Sep;105(9):1633-9. doi: 10.1111/j.1360-0443.2010.03031.x. PMID 20707781